CLINICAL TRIAL: NCT05697965
Title: TheUseofLocalVancomycinPowdertoPreventPeriprostheticJointInfectioninPrimaryTotalHipandKneeArthroplasty.ARandomizedControlledTrial.
Brief Title: LocalVancomycinPowderToPreventPeriprostheticJointInfection.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maro Maher Botros Boktor, Resident physician at Orthopedic& Trauma department,principal investigator, Assiut University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Vancomycin in Arthroplasty
Record Dates: First submitted 2022-07-12; First posted 2023-01-26 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Arthroplasty Complications; Periprosthetic Fracture of Hip
MeSH Terms: interventions — Vancomycin; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vancomycin loaded group (Experimental): applying 1 gm of vancomycin powder intracapsularly during primary total knee and hip arthroplasty operations
  Interventions: Drug: Vancomycin; Procedure: Total knee or total hip arthroplasty
- Non vancomycin loaded group (Experimental): Total knee & hip arthroplasty done without applying local vancomycin powder comparing the results with vancomycin loaded group
  Interventions: Procedure: Total knee or total hip arthroplasty

INTERVENTIONS:
Drug: Vancomycin — applying 1 gm of vancomycin powder intracapsularly during primary total knee and hip arthroplasty to prevent periprosthetic joint infection
  Other Names: Vancomycin sulphate
  Arms: Vancomycin loaded group
Procedure: Total knee or total hip arthroplasty — Primary total knee or total hip arthroplasty without using local vancomycin

SUMMARY:
The purpose of this study is to evaluate the efficacy and complication profile of local vancomycin application in primary arthroplasty. The investigators hypothesized that the use of local antibiotics would decrease the rate of infection compared to controls and this will be achieved by applying 1 gm of vancomycin powder intracapsularly.

DETAILED DESCRIPTION:
Periprosthetic joint infection is a truly devastating complication of total joint arthroplasty (TJA), causing most patients to undergo a revision surgery and to bear significant psychological and financial burden. Surveys suggest patients of total joint arthroplasty undergoing revision for infection have poorer functional outcomes and satisfaction levels than patients undergoing revision for other reasons, with negative consequences being more persistent .

Despite developments in infection prophylaxis and risk factor mitigation, patients with periprosthetic joint infection represent a substantial societal and monetary cost to our value-based health care system. Thus, there is significant interest in developing and systematically evaluating new PJI prophylaxis measures to reduce this rate.

Historically, local wound vancomycin powder has been shown to safely reduce infection rates in spine surgery. The earliest and strongest support for local vancomycin powder for primary orthopedic surgery came from the spine literature, and it now has support in the shoulder and elbow and foot and ankle literature. The use of topical vancomycin was first reported in 1989 when the application of topical vancomycin to the sternum in cardio thoracic patients reduced rates of sternal infection from 3.6% to 0.45%). Similarly, multiple studies have shown that vancomycin decreases the rate of postoperative infections in patients undergoing spinal surgery.

Importantly, data on topical vancomycin powder used alone remain inconclusive for TJA, with some stating that it may increase aseptic wound complications, and others stating that it reduces PJI significantly .

ELIGIBILITY:
Inclusion Criteria:

all patients population who will undergo primary total knee or total hip arthroplasty

Exclusion Criteria:

* patients with diabetes mellitus inflammatory arthritis diseases smokers BMI > 40

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Follow up for infected patients after 90 days with surgical site infection. | 3 months after operation
  The purpose of this study is evaluation of the efficacy and complication profile of local vancomycin application in primary arthroplasty. The use of local antibiotics would decrease the rate of infection compared to controls and this will be achieved by applying 1 gm of vancomycin powder intracapsularly that will be evaluated by inflammatory markers CRP (if more than 1 gm/dl), ESR(more than 20) as laboratory investigations.

SECONDARY OUTCOMES:
Aseptic wound complications such as skin erosion, wound dehiscence, and prolonged wound healing. | 3 months
  The purpose of this study is evaluation of the efficacy and complication profile of local vancomycin application in primary arthroplasty. The investigators hypothesized that the use of local antibiotics would decrease the rate of infection compared to controls and this will be achieved by applying 1 gm of vancomycin powder intracapsularly by examination wound site if there's surgical site infection, dehescience, abscess, discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Yossef Saleh, Principal Investigator — Vice president

REFERENCES:
- [Background] Wukich DK, Dikis JW, Monaco SJ, Strannigan K, Suder NC, Rosario BL. Topically Applied Vancomycin Powder Reduces the Rate of Surgical Site Infection in Diabetic Patients Undergoing Foot and Ankle Surgery. Foot Ankle Int. 2015 Sep;36(9):1017-24. doi: 10.1177/1071100715586567. Epub 2015 May 12. PMID 25967254
- [Background] Kurtz SM, Lau E, Watson H, Schmier JK, Parvizi J. Economic burden of periprosthetic joint infection in the United States. J Arthroplasty. 2012 Sep;27(8 Suppl):61-5.e1. doi: 10.1016/j.arth.2012.02.022. Epub 2012 May 2. PMID 22554729
- [Background] Sweet FA, Roh M, Sliva C. Intrawound application of vancomycin for prophylaxis in instrumented thoracolumbar fusions: efficacy, drug levels, and patient outcomes. Spine (Phila Pa 1976). 2011 Nov 15;36(24):2084-8. doi: 10.1097/BRS.0b013e3181ff2cb1. PMID 21304438
- [Background] Yan H, He J, Chen S, Yu S, Fan C. Intrawound application of vancomycin reduces wound infection after open release of post-traumatic stiff elbows: a retrospective comparative study. J Shoulder Elbow Surg. 2014 May;23(5):686-92. doi: 10.1016/j.jse.2014.01.049. PMID 24745317